CLINICAL TRIAL: NCT05679973
Title: Evaluation of the Efficacy of Polybutester Suture on Postoperative Complications in Lower Impacted Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, levent Cigerim, Head of Oral and Maxillofacial Surgery Department, Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 03.07.2019/11
Record Dates: First submitted 2022-02-16; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Impacted Third Molar Tooth
Keywords: Polybutester; Polypropylene; Pain; Edema; Trismus
MeSH Terms: conditions — Pain; Edema; Trismus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polybutester (Experimental): Polybutester suture is a copolymer of polyglycol terephthalate and polybutylene terephthalate. It is a synthetic, non-resorbable, monofilament suture material. Polybutester is stronger than other monofilaments. Suture memory is poor and packaging does not retain its shape. Therefore, this suture is easier to work with and the knot security is higher. Polybutester suture adapts better to tensile strength than other synthetic sutures. This suture adapts to the increasing wound edema and returns to its original shape when the edema subsides. Also, this suture reduces the risk of hypertrophic scar formation due to its ability to adapt to the edema and changing configuration of a healing wound. It produces better cosmetic results.
  Interventions: Device: Polybutester suture
- Polypropylene (Active Comparator): Polypropylene, used as suture material, is formed by bringing isotactic stereoisomers of a linear hydrocarbon crystalline polymer into sterile monofilament form. Polymer polypropylene is a non-resorbable, synthetic, monofilament suture. It has high compressive strength and low tissue reactivity. It is resistant to infection formation. In general, the ability to close and protect the wound is good. The suture memory is high, therefore it is difficult to use and the knot security is less than other sutures. Allergic reaction due to polypropylene sutures is very rare.
  Interventions: Device: Polypropylene suture

INTERVENTIONS:
Device: Polybutester suture — After third molar surgery this suture used for primary closure.
  Arms: Polybutester
Device: Polypropylene suture — After third molar surgery this suture used for primary closure.
  Arms: Polypropylene

SUMMARY:
This study aimed to evaluate the efficacy of polybutester sutures on postoperative complications in lower impacted third molar surgery.

DETAILED DESCRIPTION:
After extraction of the bilateral lower third molars (35 patients), two different types of sutures were used on each side. Group 1( Polybutester suture) , group 2 (Polypropylene suture). Measurements to evaluate edema, trismus, and pain (using the VAS scale) had been taken pre-procedure and post-procedure( 2nd and 7th day )

ELIGIBILITY:
Inclusion Criteria:

* Any medication until 2 weeks before the operations,
* Impacted teeth in mesial and horizontal positions and in class 2 and class B according to Pell & Gregory classification,
* Asymptomatic impacted teeth.
* Coming to control and fill in the given and requested forms,
* Regularly use the given drugs

Exclusion Criteria:

* Systemic disease,
* Smoking,
* Pregnancy or breastfeeding,
* Allergy to the drugs to be used in the study,
* Using any additional medication that may affect the outcome of the study,
* Post-operative alveolitis.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Pain Evaluation | Postoperative 1st day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | Postoperative 2nd day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | Postoperative 3rd day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | Postoperative 5th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | Postoperative 7th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Edema evaluation using Facial measurement | Preoperative
  The distance between predetermined facial anatomic landmarks (from the mandibular angle to lateral corner of the eye, from tragus to labial commissura, and from tragus to soft tissue pogonion) which was measured with using thread and millimeter ruler.
Edema evaluation using Facial measurement | Postoperative 2nd day
  Postoperative edema was evaluated by the distance between predetermined facial anatomic landmarks (from the mandibular angle to lateral corner of the eye, from tragus to labial commissura, and from tragus to soft tissue pogonion) which was measured with using thread and millimeter ruler.
Edema evaluation | Postoperative 7th day
  Postoperative edema was evaluated by the distance between predetermined facial anatomic landmarks (from the mandibular angle to lateral corner of the eye, from tragus to labial commissura, and from tragus to soft tissue pogonion) which was measured with using thread and millimeter ruler.
Trismus Evaluation | Preoperative
  Preoperative trismus was evaluated by the maximum distance between the incisive borders of the upper and lower right incisive teeth which were measured with a caliper.
Trismus evaluation | Postoperative 2nd day
  Postoperative trismus was evaluated by the maximum distance between the incisive borders of the upper and lower right incisive teeth which was measured with a caliper.
Trismus evaluation | Postoperative 7th day
  Postoperative trismus was evaluated by the maximum distance between the incisive borders of the upper and lower right incisive teeth which was measured with a caliper.

CONTACTS AND LOCATIONS:
Overall Officials: Levent Ciğerim, Assoc.Prof., Study Director — Yuzuncu Yil University
Locations (1):
- Van Yuzuncu Yil University, Faculty of Dentistry, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT05679973/ICF_000.pdf